CLINICAL TRIAL: NCT06123845
Title: Pressure HIgh or LOw DElivered to Preterm Newborns in the Delivery ROOM
Acronym: PHILODENDROOM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: ASST Fatebenefratelli Sacco (Other)
Responsible Party: Principal Investigator, Francesco Cavigioli, Principal Investigator, ASST Fatebenefratelli Sacco
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018//ST/231
Record Dates: First submitted 2023-10-30; First posted 2023-11-09 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Respiratory Distress Syndrome in Premature Infant
Keywords: RDS; NCPAP; PEEP; lung recruitment; delivery room resuscitation

STUDY DESIGN:
Intervention Model Description: Sealed opaque envelopes randomization
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CPAP 8 (Experimental): Upon arrival of the infant on the neonatal resuscitation trolley, start the normal standard procedures required by international protocols (e.g., drying, temperature control measures, placement of pulse-oximeter sensor to the right hand or wrist, etc.). Immediately start CPAP application with mask and T-piece: the CPAP level will be set at 8 cmH2O. Perform gentle tactile stimulation if the child is not breathing in appropriately. Place the pulse-oximeter sensor on the right hand then connect it to the oxymeter previously turned on. Assess breathing and HR for 30 seconds. Perform the next step of the flow-chart of resuscitation in the delivery room according to the Neonatal Resuscitation Program guidelines. If positive pressure ventilation (PPV) is required (in case of persistent bradycardia or apnea), maintain PEEP at 8 cm H2O and an initial PIP of 25 cm H2O. The CPAP level will be reduced to 6 cm H2O after 15 minutes of life, then the recording will be discontinued.
  Interventions: Behavioral: static CPAP 8 cmH2O
- CPAP 5 (Active Comparator): Upon arrival of the infant on the neonatal resuscitation trolley, start the normal standard procedures required by international protocols (e.g., drying, temperature control measures, placement of pulse-oximeter sensor to the right hand or wrist, etc.). Immediately start CPAP application with mask and T-piece: the CPAP level will be set at 5 cmH2O. Perform gentle tactile stimulation if the child is not breathing in appropriately. Place the pulse-oximeter sensor on the right hand then connect it to the oxymeter previously turned on. Assess breathing and HR for 30 seconds. Perform the next step of the flow-chart of resuscitation in the delivery room according to the Neonatal Resuscitation Program guidelines. If positive pressure ventilation (PPV) is required (in case of persistent bradycardia or apnea), maintain PEEP at 5 cm H2O and an initial PIP of 25 cm H2O. The CPAP level will be raised to 6 cm H2O after 15 minutes of life, then the recording will be discontinued.
  Interventions: Behavioral: static CPAP 5 cmH2O

INTERVENTIONS:
Behavioral: static CPAP 8 cmH2O — Set static CPAP or PEEP pressure level at 8 cmH2O
  Arms: CPAP 8
Behavioral: static CPAP 5 cmH2O — Set static CPAP or PEEP pressure level at 5 cmH2O
  Arms: CPAP 5

SUMMARY:
The aim of this randomized pilot clinical trial of preterm infants requiring noninvasive respiratory support for respiratory distress syndrome (RDS) at birth is to improve short-term respiratory outcomes. The main question it aims to answer is:

* Can a CPAP (or a PEEP if ventilation is needed) administered with a face mask and a T-piece at a level of 8 cmH2O improve lung recruitment in the delivery room when compared to administration of a level of 5 cmH2O in a control group?
* Secondly, can improved lung recruitment in the first few minutes of life provide long-term benefits to the premature infant? The participants will be premature infants between 26 and 29+6 weeks gestational age.

DETAILED DESCRIPTION:
BACKGROUND:

It has been widely demonstrated that noninvasive respiratory support (NIV) used in the delivery room can reduce the incidence of pulmonary bronchodysplasia (BPD) and death in very preterm infants weighting less than 1500 g.

In this population, the use of CPAP immediately after birth during the respiratory stabilization in the delivery room has been shown to promote respiratory transition and promote the achievement of an initial adequate functional residual capacity (CFR).

To date, various forms of delivery of additional pressures in the first minutes of life are being studied such as positive pressure ventilation (PPV), sustained inflation (SI), ventilation with dynamic increasing and decreasing levels of CPAP. However, there is no consensus on which pressure is the best and safest to apply and its optimal duration.

This monocentric pilot study aims to verify in preterm infants (26-29+6 weeks EG) the feasibility, efficacy and safety of using two different levels of CPAP (5 vs 8 cmH2O - both of which are contemplated in international guidelines for the management of the premature infant) in the delivery room; it will also test the accuracy and usefulness of the data that can be recorded with an RFM as indices of oxygenation, spontaneous ventilation and therefore of early lung recruitment. The investigators hypothesize that a higher CPAP level (8 cmH2O) for the first 15 minutes of life may lead to faster and more effective lung recruitment.

Statistical calculation The investigators use, as an index of early lung recruitment and as the primary outcome of the study, the SpO2/FiO2 (S/F) ratio as reported in the literature. The investigators calculated that the mean of this value at the end of the early phase of lung recruitment in the delivery room, in an historical local population of premature infants is 271+/-140. Wanting to improve this ratio, and thinking that it is possible to bring it to an average value of 316, (this goal can be achieved by reducing the need for Oxygen in the DR by about 0.05), it was calculated that with alpha=0.05 and beta=0.20 (study power of 80%), the number of patients to be enrolled is equal to 152 infants for each of the two main arms of the study. Given the large size of the sample, for which the involvement of numerous Level III neonatology centers, the investigators considered appropriate to undertake a pilot study to verify its feasibility, enrollment time, costs and moreover to assess and verify proper monitoring with a respiratory Function Monitor (RFM) and the possibility to improve the assessment of primary and secondary outcomes in the final large-scale designed study. To calculate the sample size of the pilot study, the investigators applied the method of calculation described and published by Cocks T. et al in 2013, considering an upper confidence limit of 90%. It was calculated an enrollment of a total of 56 infants (18% of the main study's sample size), or 28 infants for each of the two arms of the study.

In the investigator's Neonatologic Center a maximum of 20 patients per year could realistically be enrolled. It was therefore necessary to involve other centers in this study that had equally the ability and experience in using this equipments in the delivery room. A Neonatal Intensive Care Unit in Canada, which had initially given willingness to participate in the study was later on stopped because of the occurrence of the covid pandemic. Other centers may be involved at a later date for the main study.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants at birth between 26 and 29+6 weeks gestational age with Respiratory distress syndrome requiring non invasive respiratory support

Exclusion Criteria:

* Congenital anomalies

Ages: 26 Weeks to 30 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Estimated)
Dates: Start 2019-04-11 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Oxygen saturation/Inspired Oxygen fraction (SpO2/FiO2) | From randomization assessed every minute up to 15 minutes of life
  Oxygen saturation / Inspired Oxygen fraction ratio

SECONDARY OUTCOMES:
Exhaled tidal volumes (Vte) | From randomization assessed every minute up to 15 minutes of life
  Exhaled tidal volumes
HR | From randomization assessed every minute up to 15 minutes of life
  Heart rate
SpO2 | From randomization assessed every minute up to 15 minutes of life
  Oxygen peripheral saturation
PPV | From randomization up to 15 minutes of life
  Need for positive pressure ventilation
ET | From randomization up to 15 minutes of life
  occurrence of Endotracheal intubation in the delivery room
MV | From randomization up to 72 hours of life
  Need for Mechanical ventilation
Surf | From randomization up to 72 hours of life
  Need for Surfactant administration
PNX | From randomization up to 72 hours of life
  occurrence of Pneumothorax
PIE | From randomization up to 72 hours of life
  occurrence of Pulmonary interstitial emphysema
IVH | From randomization up to 72 hours of life
  occurrence of Intraventricular hemorrhage any grade of severity
BPD | assessed at 36 weeks gestational age (GA)
  Clinical diagnosis of Bronchopulmonary dysplasia
Death | From date of randomization until the date of death from any cause, assessed up to 40 weeks gestational age (GA)
  Mortality for any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale dei Bambini Vittore Buzzi, Milan, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No
A database of participants' blacked-out names will be shared with statisticians for analysis